CLINICAL TRIAL: NCT02943330
Title: Relation Between Depression, Genes, Cytokines, Chronic Fatigue, Physical Illnesses and Quality of Life
Brief Title: Depression, Genes, Cytokines, Chronic Fatigue, Physical Illnesses and Quality of Life
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chih-Ken Chen, Professor, Chang Gung Memorial Hospital
Other Study IDs: 98-2314-B-182-023-MY3
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Hemodialysis; Hepatitis C
Keywords: Depression; Cytokines; Hemodialysis; Interferon treatment; Hepatitis C
MeSH Terms: conditions — Hepatitis C; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — IL-1β, IL-6 and TNF-α, as well as genotype the 5-HTTLPR triallelic polymorphism on all subjects.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodialysis: Hemodialysis patients
  Interventions: Other: Questionnaire
- Hepatitis C: Patients receiving interferon treatment for hepatitis C
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaires such as Hospital Anxiety and Depression Scale (HADS) and Montgomery Asberg Depression Rating Scale (MADRS), Short-form Health-related Quality of Life (SF-36), as well as psychiatric diagnostic interview with the Mini-International Neuropsychiatric Interview (MINI) and the Family Interview for Genetic Study (FIGS).

SUMMARY:
Depression is one of the most common psychiatric diseases, with prevalence estimates ranging from 5% to 20%. Depression is now recognized as a brain disease; it can be managed and treated effectively with a wide range of options, but its biological basis is still far from clear. Studies of monozygotic and dizygotic twin pairs suggest polygenic inheritance, with an overall heritability estimate between 40% and 70 %. Gene-environment interaction has been recognized for a long time in the pathophysiology of depression, and its best biological substratum at present is represented by the serotonin transporter (5-HTT) gene. It would be interesting to study association between the novel allelic variants or at least the triallelic 5-HTTLPR polymorphism and depression. Depression is common in patients with end-stage renal disease and to occur in about 20% to 30% of hemodialysis patients. Interferon-induced depression is estimated up to 50% among patients with hepatitis C. Several sets of observations support the supposition that cytokines, and proinflammatory cytokines in particular, are involved in depressive disorders. Depression sufferers have been reported to have elevated blood levels of interleukin 1 (IL-1), IL-6 and tumor necrosis factor α (TNF-α).

DETAILED DESCRIPTION:
The aim of this study is to examine the relations between depression and psychiatric family history, candidate genes, cytokines and health-related quality of life among hemodialysis patients and patients receiving interferon treatment for hepatitis C. The investigators aim to recruit 200 hemodialysis patients and 100 patients receiving interferon treatment for hepatitis C at Chang Gung Memorial Hospital, Keelung. Our pilot study found that among hemodialysis patients, the prevalence rates of probable anxiety disorder and probably depression disorder was 25.9% and 40.0%. Among the patients receiving interferon treatment for hepatitis C, the prevalence rates of probable anxiety disorder and probably depression disorder was 30.2% and 20.7% at baseline, and 44.0% and 36.2% at 3 months after interferon treatment. The study procedure consists of 2 parts. For the first one, all the recruited hemodialysis patients will receive assessments for fatigue symptoms using Fatigue Scale, depressive symptoms using Hospital Anxiety and Depression Scale (HADS) and Montgomery Asberg Depression Rating Scale (MADRS), Short-form Health-related Quality of Life (SF-36), blood levels of IL-1β, IL-6 and TNF-αas well as psychiatric diagnostic interview with the Mini-International Neuropsychiatric Interview (MINI) and the Family Interview for Genetic Study (FIGS). The second one is a prospective follow up of patients receiving interferon treatment. Before initiating interferon treatment, the subjects will receive baseline assessments using the same scales mentioned above. The investigators will genotype the 5-HTTLPR triallelic polymorphism on all subjects. The follow-up visits are at month 1, month 3, termination, and one month after termination of interferon program. This proposed project will provide a broad view and better understanding of the gene-environment interaction in the etiology of depression.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or more, both males and females
* Agree to participate and able to write Informed consent.

Exclusion Criteria:

* No specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to recruit 200 demodialysis patients and 100 patients receiving interferon treatment for hepatitis C at Chang Gung Memorial Hospital, Keelung.
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Psychiatric diagnosis | 3 years
  Psychiatric diagnosis will be made according to DSM IV criteria after a structured psychiatric diagnosis interview with the Mini-International Neuropsychiatric Interview (MINI).

SECONDARY OUTCOMES:
Psychiatric family history | 3 years
  Psychiatric family history will be obtained by interviewing with the Chinese version of the Diagnostic Interview for Genetic Study. Based on the informant's responses to the general screening questions, five symptom checklists (depression, mania, alcohol and other drug abuse, psychosis, paranoid/schizoid/ schizotypal personality disorder) were completed for each first-degree relative.
Hospital Anxiety and Depression Scale | 3 years
  Depressive symptoms will be evaluated using Hospital Anxiety and Depression Scale (HADS) and Montgomery Asberg Depression Rating Scale (MADRS). The HADS is a self-reported scale, and consists of 14 items (7 for anxiety and 7 for depression), which has been frequently applied to assess anxiety and depression symptoms of medically ill patients.
Montgomery Asberg Depression Rating Scale | 3 years
  The MADRS is a rating scale for severity of depressive mood symptoms. The scale consists of 10 items. Each item is rated from 0 to 6. The MADRS total score is the sum of the 10 items, and the score ranges from 0 to 60.
Quality of life | 3 years
  Quality of life will be assessed using the Short-form Health-related Quality of Life (SF-36) . This questionnaire assesses eight dimensions of physical and mental health, and the range is from 100 (optimal) to zero (poorest): physical functioning, physical role functioning, bodily pain, general health, vitality, social functioning, emotional role functioning, and mental health.
  The SF-36 has demonstrated sensitivity to change, and score changes can be interpreted as changes in the health-related quality of life of the patient.
Fatigue symptoms | 3 years
  Fatigue symptoms will be evaluated using the self-reported Fatigue Scale.
Cytokines | 3 years
  The levels of interleukin 1, interleukin 6, tumor necrosis factor α, DHEA, and DHEA-S will be tested via standard ELISA protocol.
Genotyping | 3 years
  The Genomic DNA will be extracted from peripheral blood by standard methods.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Ken Chen, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beck AT, Steer RA, Kovacs M, Garrison B. Hopelessness and eventual suicide: a 10-year prospective study of patients hospitalized with suicidal ideation. Am J Psychiatry. 1985 May;142(5):559-63. doi: 10.1176/ajp.142.5.559. PMID 3985195
- [Result] Cadoret RJ. Evidence for genetic inheritance of primary affective disorder in adoptees. Am J Psychiatry. 1978 Apr;135(4):463-6. doi: 10.1176/ajp.135.4.463. PMID 637144
- [Result] Campi-Azevedo AC, Boson W, De Marco L, Romano-Silva MA, Correa H. Association of the serotonin transporter promoter polymorphism with suicidal behavior. Mol Psychiatry. 2003 Nov;8(11):899-900. doi: 10.1038/sj.mp.4001381. No abstract available. PMID 14593426
- [Result] Capuron L, Miller AH. Cytokines and psychopathology: lessons from interferon-alpha. Biol Psychiatry. 2004 Dec 1;56(11):819-24. doi: 10.1016/j.biopsych.2004.02.009. PMID 15576057
- [Result] Caspi A, Sugden K, Moffitt TE, Taylor A, Craig IW, Harrington H, McClay J, Mill J, Martin J, Braithwaite A, Poulton R. Influence of life stress on depression: moderation by a polymorphism in the 5-HTT gene. Science. 2003 Jul 18;301(5631):386-9. doi: 10.1126/science.1083968. PMID 12869766
- [Result] Chalder T, Berelowitz G, Pawlikowska T, Watts L, Wessely S, Wright D, Wallace EP. Development of a fatigue scale. J Psychosom Res. 1993;37(2):147-53. doi: 10.1016/0022-3999(93)90081-p. PMID 8463991
- [Result] Chen WJ, Liu SK, Chang CJ, Lien YJ, Chang YH, Hwu HG. Sustained attention deficit and schizotypal personality features in nonpsychotic relatives of schizophrenic patients. Am J Psychiatry. 1998 Sep;155(9):1214-20. doi: 10.1176/ajp.155.9.1214. PMID 9734545
- [Result] Chisholm D, Sanderson K, Ayuso-Mateos JL, Saxena S. Reducing the global burden of depression: population-level analysis of intervention cost-effectiveness in 14 world regions. Br J Psychiatry. 2004 May;184:393-403. doi: 10.1192/bjp.184.5.393. PMID 15123502
- [Result] Chou FH, Chou P, Su TT, Ou-Yang WC, Chien IC, Lu MK, Huang MW. Quality of life and related risk factors in a Taiwanese Village population 21 months after an earthquake. Aust N Z J Psychiatry. 2004 May;38(5):358-64. doi: 10.1080/j.1440-1614.2004.01364.x. PMID 15144515
- [Result] Gershon ES, Hamovit J, Guroff JJ, Dibble E, Leckman JF, Sceery W, Targum SD, Nurnberger JI Jr, Goldin LR, Bunney WE Jr. A family study of schizoaffective, bipolar I, bipolar II, unipolar, and normal control probands. Arch Gen Psychiatry. 1982 Oct;39(10):1157-67. doi: 10.1001/archpsyc.1982.04290100031006. PMID 7125846
- [Result] Goldney RD, Fisher LJ, Wilson DH, Cheok F. Suicidal ideation and health-related quality of life in the community. Med J Aust. 2001 Nov 19;175(10):546-9. doi: 10.5694/j.1326-5377.2001.tb143717.x. PMID 11795547
- [Result] Heils A, Teufel A, Petri S, Stober G, Riederer P, Bengel D, Lesch KP. Allelic variation of human serotonin transporter gene expression. J Neurochem. 1996 Jun;66(6):2621-4. doi: 10.1046/j.1471-4159.1996.66062621.x. PMID 8632190
- [Result] Hestad KA, Tonseth S, Stoen CD, Ueland T, Aukrust P. Raised plasma levels of tumor necrosis factor alpha in patients with depression: normalization during electroconvulsive therapy. J ECT. 2003 Dec;19(4):183-8. doi: 10.1097/00124509-200312000-00002. PMID 14657769
- [Result] Horsmans Y. Interferon-induced depression in chronic hepatitis C. J Antimicrob Chemother. 2006 Oct;58(4):711-3. doi: 10.1093/jac/dkl331. Epub 2006 Sep 2. PMID 16951413
- [Result] Hu XZ, Lipsky RH, Zhu G, Akhtar LA, Taubman J, Greenberg BD, Xu K, Arnold PD, Richter MA, Kennedy JL, Murphy DL, Goldman D. Serotonin transporter promoter gain-of-function genotypes are linked to obsessive-compulsive disorder. Am J Hum Genet. 2006 May;78(5):815-826. doi: 10.1086/503850. Epub 2006 Mar 28. PMID 16642437
- [Result] Kelley KW, Bluthe RM, Dantzer R, Zhou JH, Shen WH, Johnson RW, Broussard SR. Cytokine-induced sickness behavior. Brain Behav Immun. 2003 Feb;17 Suppl 1:S112-8. doi: 10.1016/s0889-1591(02)00077-6. PMID 12615196
- [Result] Kuo CJ, Tang HS, Tsay CJ, Lin SK, Hu WH, Chen CC. Prevalence of psychiatric disorders among bereaved survivors of a disastrous earthquake in taiwan. Psychiatr Serv. 2003 Feb;54(2):249-51. doi: 10.1176/appi.ps.54.2.249. PMID 12556609
- [Result] Kuo WH, Gallo JJ, Tien AY. Incidence of suicide ideation and attempts in adults: the 13-year follow-up of a community sample in Baltimore, Maryland. Psychol Med. 2001 Oct;31(7):1181-91. doi: 10.1017/s0033291701004482. PMID 11681544
- [Result] Lesch KP, Gutknecht L. Pharmacogenetics of the serotonin transporter. Prog Neuropsychopharmacol Biol Psychiatry. 2005 Jul;29(6):1062-73. doi: 10.1016/j.pnpbp.2005.03.012. PMID 15951088
- [Result] Maes M, Vandoolaeghe E, Ranjan R, Bosmans E, Bergmans R, Desnyder R. Increased serum interleukin-1-receptor-antagonist concentrations in major depression. J Affect Disord. 1995 Dec 24;36(1-2):29-36. doi: 10.1016/0165-0327(95)00049-6. PMID 8988262
- [Result] Mendlewicz J, Rainer JD. Adoption study supporting genetic transmission in manic--depressive illness. Nature. 1977 Jul 28;268(5618):327-9. doi: 10.1038/268327a0. No abstract available. PMID 887159
- [Result] Miller DB, O'Callaghan JP. Depression, cytokines, and glial function. Metabolism. 2005 May;54(5 Suppl 1):33-8. doi: 10.1016/j.metabol.2005.01.011. PMID 15877311
- [Result] Nakamura M, Ueno S, Sano A, Tanabe H. The human serotonin transporter gene linked polymorphism (5-HTTLPR) shows ten novel allelic variants. Mol Psychiatry. 2000 Jan;5(1):32-8. doi: 10.1038/sj.mp.4000698. PMID 10673766
- [Result] Nascimento I, Nardi AE, Valenca AM, Lopes FL, Mezzasalma MA, Nascentes R, Zin WA. Psychiatric disorders in asthmatic outpatients. Psychiatry Res. 2002 May 15;110(1):73-80. doi: 10.1016/s0165-1781(02)00029-x. PMID 12007595
- [Result] Nurnberger JI Jr, Blehar MC, Kaufmann CA, York-Cooler C, Simpson SG, Harkavy-Friedman J, Severe JB, Malaspina D, Reich T. Diagnostic interview for genetic studies. Rationale, unique features, and training. NIMH Genetics Initiative. Arch Gen Psychiatry. 1994 Nov;51(11):849-59; discussion 863-4. doi: 10.1001/archpsyc.1994.03950110009002. PMID 7944874
- [Result] Perlman RL, Finkelstein FO, Liu L, Roys E, Kiser M, Eisele G, Burrows-Hudson S, Messana JM, Levin N, Rajagopalan S, Port FK, Wolfe RA, Saran R. Quality of life in chronic kidney disease (CKD): a cross-sectional analysis in the Renal Research Institute-CKD study. Am J Kidney Dis. 2005 Apr;45(4):658-66. doi: 10.1053/j.ajkd.2004.12.021. PMID 15806468
- [Result] Pirkis J, Burgess P, Dunt D. Suicidal ideation and suicide attempts among Australian adults. Crisis. 2000;21(1):16-25. doi: 10.1027//0227-5910.21.1.16. PMID 10793467
- [Result] Ritchie K, Artero S, Beluche I, Ancelin ML, Mann A, Dupuy AM, Malafosse A, Boulenger JP. Prevalence of DSM-IV psychiatric disorder in the French elderly population. Br J Psychiatry. 2004 Feb;184:147-52. doi: 10.1192/bjp.184.2.147. PMID 14754827
- [Result] Sakai K, Nakamura M, Ueno S, Sano A, Sakai N, Shirai Y, Saito N. The silencer activity of the novel human serotonin transporter linked polymorphic regions. Neurosci Lett. 2002 Jul 12;327(1):13-6. doi: 10.1016/s0304-3940(02)00348-8. PMID 12098489
- [Result] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Result] Simon GE, Von Korff M, Lin E. Clinical and functional outcomes of depression treatment in patients with and without chronic medical illness. Psychol Med. 2005 Feb;35(2):271-9. doi: 10.1017/s0033291704003071. PMID 15841684
- [Result] Sullivan PF, Neale MC, Kendler KS. Genetic epidemiology of major depression: review and meta-analysis. Am J Psychiatry. 2000 Oct;157(10):1552-62. doi: 10.1176/appi.ajp.157.10.1552. PMID 11007705
- [Result] Suominen K, Isometsa E, Suokas J, Haukka J, Achte K, Lonnqvist J. Completed suicide after a suicide attempt: a 37-year follow-up study. Am J Psychiatry. 2004 Mar;161(3):562-3. doi: 10.1176/appi.ajp.161.3.562. PMID 14992984
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Result] Weissman MM, Bland RC, Canino GJ, Greenwald S, Hwu HG, Joyce PR, Karam EG, Lee CK, Lellouch J, Lepine JP, Newman SC, Rubio-Stipec M, Wells JE, Wickramaratne PJ, Wittchen HU, Yeh EK. Prevalence of suicide ideation and suicide attempts in nine countries. Psychol Med. 1999 Jan;29(1):9-17. doi: 10.1017/s0033291798007867. PMID 10077289
- [Result] Weissman MM, Gershon ES, Kidd KK, Prusoff BA, Leckman JF, Dibble E, Hamovit J, Thompson WD, Pauls DL, Guroff JJ. Psychiatric disorders in the relatives of probands with affective disorders. The Yale University--National Institute of Mental Health Collaborative Study. Arch Gen Psychiatry. 1984 Jan;41(1):13-21. doi: 10.1001/archpsyc.1984.01790120015003. PMID 6691780
- [Result] Wender PH, Kety SS, Rosenthal D, Schulsinger F, Ortmann J, Lunde I. Psychiatric disorders in the biological and adoptive families of adopted individuals with affective disorders. Arch Gen Psychiatry. 1986 Oct;43(10):923-9. doi: 10.1001/archpsyc.1986.01800100013003. PMID 3753159
- [Result] Yang SC, Kuo PW, Wang JD, Lin MI, Su S. Quality of life and its determinants of hemodialysis patients in Taiwan measured with WHOQOL-BREF(TW). Am J Kidney Dis. 2005 Oct;46(4):635-41. doi: 10.1053/j.ajkd.2005.06.015. PMID 16183418
- [Derived] Wang LJ, Chen SW, Chen CK, Yen CL, Chang JJ, Lee TS, Liu CJ, Chen LW, Chien RN. Treatment-emergent depression and anxiety between peginterferon alpha-2a versus alpha-2b plus ribavirin for chronic hepatitis C. BMC Psychiatry. 2016 Nov 25;16(1):424. doi: 10.1186/s12888-016-1135-8. PMID 27884134